CLINICAL TRIAL: NCT04207398
Title: TIPS vs. NSBB Plus Endotherapy for the Prevention of Variceal Rebleeding in NSBB Non-responders of Primary Prophylaxis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Tie Jun, Director of clinical research, Air Force Military Medical University, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KY20192149-C-1
Record Dates: First submitted 2019-11-27; First posted 2019-12-20 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Variceal Hemorrhage; TIPS; NSBB; Liver Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis | interventions — Combined Modality Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TIPS (Experimental): Transjugular intrahepatic portosystemic shunt (TIPS) is a procedure that uses imaging guidance to connect the portal vein to the hepatic vein in the liver.
  Interventions: Procedure: Transjugular intrahepatic portosystemic shunts
- NSBB+EBL (Active Comparator): Participants randomized to this group will receive the combination therapy of non-selective beta-blocker (NSBB) and endoscopic band ligation (EBL) . NSBB, including propranolol and carvidilol, will be started at day 5 after the index bleeding and elective EBL sessions started 2 weeks after the index bleeding.
  Interventions: Other: Nonselective β-blocker (NSBB)+ endoscopic band ligation (EBL)

INTERVENTIONS:
Procedure: Transjugular intrahepatic portosystemic shunts — Transjugular intrahepatic portosystemic shunt (TIPS) is a procedure that uses imaging guidance to connect the portal vein to the hepatic vein in the liver. A small metal device called a stent is placed to keep the connection open and allow it to bring blood draining from the bowel back to the heart. TIPS may successfully reduce internal bleeding in the stomach and esophagus in patients with cirrhosis and may also reduce the accumulation of fluid in the abdomen (ascites).
  Arms: TIPS
Other: Nonselective β-blocker (NSBB)+ endoscopic band ligation (EBL) — Combination therapy of nonselective β-blocker (NSBB) and endoscopic variceal ligation (EBL) will be used for participants in this group. NSBB, which will be titrated to the maximum tolerated dose aiming to decrease the heart rate by 25%, with a lower limit of 50 beats per minute, was started at day 5 after the index bleeding, unless a contraindication was present (severe arrhythmia, severe obstructive chronic obstructive pulmonary disease, or known intolerance). Endoscopic variceal ligation sessions started 2 weeks after the index bleeding and were performed every 2-4 weeks thereafter until eradication of varices, followed by endoscopic surveillance and retreatment, if indicated, every 6-12 months.
  Other Names: Combination therapy
  Arms: NSBB+EBL

SUMMARY:
Variceal bleeding (VB) is a life-threatening complication of cirrhosis with a 6-week mortality of approximately 15%-20%. The 1-year rate of recurrent VB is approximately 60% in patients without prophylaxis treatment. Therefore, all patients who survive VB must receive active treatments to prevent rebleeding. Usually, these patients are submitted to rebleeding prophylaxis with endoscopic band ligation (EBL) combined with non-selective beta-blockers (NSBB). Transjugular intrahepatic portosystemic shunts (TIPS) are reserved for those who failed endoscopic plus medical treatment.

A recent meta-analysis comparing combination therapy to monotherapy with EBL or drug therapy has demonstrated that combination therapy is only marginally more effective than NSBB alone. This suggests that NSBB is the cornerstone of combination therapy. The lowest rebleeding rates are observed in patients on secondary prophylaxis who are hepatic venous pressure gradient (HVPG) responders (defined as a reduction in HVPG below 12 mm Hg or > 20% from baseline). A recent study demonstrated that patients who have their first episode of variceal bleeding while on primary prophylaxis with NSBB have an increased risk of further bleeding and death, despite adding EBL. These patients possibly require alternative treatment approaches, such as TIPS.

The aim of the present study was to compare the effect of TIPS vs. EBL + NSBB for the prevention of rebleeding in NSBB non-responder for primary prophylaxis.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of liver cirrhosis
* Standard NSBB therapy was used for primary prophylaxis
* At least 5 days after index variceal bleeding
* Child-Pugh score <13, Model for end-stage liver disease score < 19

Exclusion Criteria:

* Gastric variceal bleeding (GOV2，IGV1，IGV2)
* History of shunt surgery
* Degree of portal vein thrombosis > 50%
* Refractory ascites
* Budd-Chiari syndrome
* Hepatocellular carcinoma or other malignant tumors
* Uncontrolled infection
* HIV
* Pregnant or breast-feeding woman
* Poor compliance

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Cumulative incidence of clinically significant variceal rebleeding | 12 months
  Recurrent melena or hematemesis resulting in either hospital admission, blood transfusion, drop in hemoglobin of at least 3 g/L, or death within 6 weeks after rebleeding.

SECONDARY OUTCOMES:
Cumulative incidence of variceal bleeding related mortality | 12 months
  Death due to variceal bleeding
Cumulative incidence of all cause mortality | 12 months
  Including liver related and non-liver related death
Cumulative incidence of hepatic encephalopathy (HE) | 12 months
  HE was evaluated and classified according to West-Haven criteria
Cumulative incidence of adverse events (AE) | 12 months
  All kinds of adverse events

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] de Souza AR, La Mura V, Reverter E, Seijo S, Berzigotti A, Ashkenazi E, Garcia-Pagan JC, Abraldes JG, Bosch J. Patients whose first episode of bleeding occurs while taking a beta-blocker have high long-term risks of rebleeding and death. Clin Gastroenterol Hepatol. 2012 Jun;10(6):670-6; quiz e58. doi: 10.1016/j.cgh.2012.02.011. Epub 2012 Feb 22. PMID 22366180